CLINICAL TRIAL: NCT05523687
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, Excretion of [14C]-PC14586 Following a Single Oral Dose in Healthy Male Participants
Brief Title: AME Study of [14C]-PC14586 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PMV Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PMV-586-103
Record Dates: First submitted 2022-08-22; First posted 2022-08-31 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Healthy Male Volunteers
Keywords: Y220C; PC14586; PMV Pharma; PMV; AME

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single, oral dose of [14C]-PC14586 (Experimental): Healthy, male participants will receive a single, oral dose of [14C]-PC14586
  Interventions: Drug: [14C]-PC14586

INTERVENTIONS:
Drug: [14C]-PC14586 — Single, oral dose of [14C]-PC14586

SUMMARY:
This study will assess the PK and rates of elimination and mass balance of total radioactivity from [14C]-PC14586

DETAILED DESCRIPTION:
PC14586 is a first-in-class, oral, small molecule p53 reactivator that is selective for the TP53 Y220C mutation. The study will assess the PK, absorption, metabolism, and excretion of [14C]-PC14586 following a single dose in healthy male participants.

The aim is to recruit approximately 8 participants with a minimum number of 6 evaluable participants.

Each participant will be admitted to the study site pre-dose on Day -1 and will remain at the study site until at least Day 14. Participants will receive a single administration of [14C]-PC14586 as oral capsules on Day 1. During this study, whole blood, plasma, urine, feces, and vomit samples (if presented) will be collected at various timepoints to characterize the absorption, metabolism, excretion, and PK of [14C]-PC14586.

The duration of the residential period will be evaluated following the administration of [14C]-PC14586 and may be extended to ensure recovery of at least 90% of the total radioactivity, or until less than 1% of dose is recovered in urine and/or feces.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking males of any race, between 18 and 55 years of age, with BMI between 18.0 and 32.0 kg/m2 inclusive.
2. In good health, determined by no clinically significant findings from medical history and evaluations at screening and check-in as assessed by the investigator.
3. Agree to use a highly effective method of contraception from check-in through 90 days after discharge.
4. History of a minimum of 1 bowel movement per day.
5. Creatinine clearance ≥90 mL/min determined using the Cockcroft-Gault equation.
6. Able to swallow capsules.

Exclusion Criteria:

1. Significant history or clinical manifestation of any medical condition, disease or disorder, as determined by the investigator.
2. Blood pressure >140 mm systolic or >90 diastolic at screening or Day -1.
3. Positive hepatitis panel and/or positive human immunodeficiency virus test
4. Use or intend to use any prescription and/or nonprescription medications/products within14 days prior to check-in.
5. Participation in a clinical study involving last administration of an investigational drug within the past 30 days prior to dosing, or within 5 half-lives of the IMP, whichever is longer, or who have participated in more than 3 radiolabeled drug studies in the last 12 months.
6. Participants who have previously completed or withdrawn from this study or any other study investigating PC14586, or have previously received PC14586.
7. Participants with a history of alcoholism or drug/chemical abuse within 2 years prior to check-in, use of tobacco or nicotine-containing products within 3 months prior to check-in or with a positive drug and/or alcohol test result at check-in.
8. A positive p53 Y220C germline test at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Characterize Maximum Plasma Concentration (Cmax) of PC14586 and PC14586 metabolite M1 (PC16163). | 1 month
  Determine Cmax for PC14586 and PC16163 in plasma.
Characterize Time to Maximum Plasma Concentration (tmax) of PC14586 and PC14586 metabolite M1 (PC16163). | 1 month
  Determine tmax for PC14586 and PC16163 in plasma.
Characterize Total Drug Exposure (AUC0-inf) of PC14586 and PC14586 metabolite M1 (PC16163). | 1 month
  Determine AUC0-inf for PC14586 and PC16163 in plasma.
Characterize Total Drug Exposure to the last measurable concentration (AUC0-t) of PC14586 and PC14586 metabolite M1 (PC16163). | 1 month
  Determine AUC0-t for PC14586 and PC16163 in plasma.
Characterize the Half-Life (t 1/2) of PC14586 and PC14586 metabolite M1 (PC16163). | 1 month
  Determine t 1/2 for PC14586 and PC16163 in plasma.
Characterize the Clearance (CL/F) of PC14586 and PC14586 metabolite M1 (PC16163) after oral administration. | 1 month
  Determine CL/F for PC14586 and PC16163 in plasma.
Characterize the Volume of Distribution (Vd/F) of PC14586 and PC14586 metabolite M1 (PC16163) after oral administration. | 1 month
  Determine Vd/F for PC14586 and PC16163 in plasma.
Determine the total radioactivity in whole blood and plasma of PC14586 and PC14586 metabolite M1 (PC16163). | 1 month
  Determine total radioactivity for PC14586 and PC16163 in whole blood and plasma.
Characterize total radioactivity (Xlast, feces) of PC14586 excreted in feces. | 1 month
  Determine total radioactivity of PC14586 excreted in feces
Characterize the half life of total radioactivity (Xt1-t2, feces) of PC14586 excreted in feces. | 1 month
  Determine half life of total radioactivity of PC14586 excreted in feces.
Characterize the fraction excreted of total radioactivity (fe last, feces) of PC14586 in feces. | 1 month
  Determine the fraction excreted of total radioactivity of PC14586 in feces.
Characterize the half-life of fraction excreted of total radioactivity (fe t1-t2, feces) of PC14586 in feces. | 1 month
  Determine half-life of fraction excreted of total radioactivity of PC14586 in feces.
Characterize total radioactivity (Xlast, urine) of PC14586 excreted in urine. | 1 month
  Determine total radioactivity of PC14586 excreted in urine.
Characterize the half life of total radioactivity (Xt1-t2, urine) of PC14586 excreted in urine. | 1 month
  Determine half life of total radioactivity of PC14586 excreted in urine.
Characterize the fraction excreted of total radioactivity (fe last, urine) of PC14586 in urine. | 1 month
  Determine the fraction excreted of total radioactivity of PC14586 in urine.
Characterize the half-life of fraction excreted of total radioactivity (fe t1-t2, urine) of PC14586 in urine. | 1 month
  Determine half-life of fraction excreted of total radioactivity of PC14586 in urine.
Characterize the renal clearance (CLr) of PC14586 in urine. | 1 month
  Determine the renal clearance of PC14586 in urine.

SECONDARY OUTCOMES:
Identification of PC14586 metabolite profiles in plasma, urine and feces. | 1 month
  Identification of PC14586 metabolites in plasma (>10% relative total drug related exposure) and excreta (>10% of excreted dose).
Identification of the incidence and severity of adverse events after administration of PC14586. | 1 month
  Number of participants with adverse events.
Identification of the incidence of laboratory abnormalities based on hematology, clinical chemistry and urine test results of PC14586. | 1 month
  Number of participants with an incidence of laboratory abnormalities in test results.
Identification of 12-lead electrocardiogram (ECG) abnormalities after a single dose of PC14586. | 1 month
  Number of participants with abnormal 12-lead ECG results.
Identification of abnormal blood pressure after a single dose of PC14586. | 1 month
  Number of participants with abnormal blood pressure.
Identification of abnormal pulse rate after a single dose of PC14586. | 1 month
  Number of participants with abnormal pulse rate.
Identification of abnormal oral body temperature after a single dose of PC14586. | 1 month
  Number of participants with abnormal oral body temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No